CLINICAL TRIAL: NCT05101356
Title: A Phase 1/2 Open Label Study of LabVax 3(22)-23 and Adjuvant GM-CSF Alone or in Combination With Pembrolizumab in Subjects With Labyrinthin-Positive Adenocarcinomas
Brief Title: A Cancer Vaccine (Labvax 3(22)-23) and GM-CSF Alone or in Combination With Pembrolizumab for the Treatment of Advanced Stage Adenocarcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianhong Li (Other)
Collaborators: National Cancer Institute (NCI) (NIH); LabyRx Immunologic Therapeutics (Unknown)
Responsible Party: Sponsor-Investigator, Tianhong Li, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#296; NCI-2021-10667 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#296 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Advanced Adenocarcinoma; Advanced Malignant Solid Neoplasm; Metastatic Adenocarcinoma; Metastatic Malignant Solid Neoplasm; Recurrent Adenocarcinoma; Recurrent Malignant Solid Neoplasm
MeSH Terms: conditions — Adenocarcinoma; Neoplasm Metastasis | interventions — Cancer Vaccines; sargramostim; Colony-Stimulating Factors; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 Treatment (sargramostim, LabVax 3(22)-23) (Experimental): Patients receive sargramostim SC and LabVax 3(22)-23 ID on weeks 1, 2, 4, 8, and 12 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Antineoplastic Vaccine; Biological: Sargramostim
- Phase 2 Treatment (sargramostim, LabVax 3(22)-23, pembrolizumab) (Experimental): Pembrolizumab will be given intravenously every 3 weeks for up to 12 cycles on Day 1 of Weeks 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 31, and 34. Participants will be given LabVax 3(22)-23 (intradermally) and adjuvant GM-CSF (subcutaneously) on weeks 7, 8, 10, 14, and 18.
  Interventions: Biological: Antineoplastic Vaccine; Biological: Sargramostim; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Antineoplastic Vaccine — Given LabVax 3(22)-23 ID
  Other Names: cancer treatment vaccine; Cancer Vaccine; Neoplasm Vaccine; Tumor Vaccine
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
Biological: Pembrolizumab — Given IV per standard of care
  Other Names: KEYTRUDA; MK-3475
  Arms: Phase 2 Treatment (sargramostim, LabVax 3(22)-23, pembrolizumab)

SUMMARY:
This phase 1/2 trial tests the safety and effectiveness of a cancer vaccine called Labvax 3(22)-23 and GM-CSF alone or in combination with pembrolizumab in treating adenocarcinoma that has spread to other places in the body (advanced stage). Labvax 3(22)-23 is designed to target a specific antigen (labyrinthin), which is a protein found on the surface of adenocarcinoma tumor cells. Labyrinthin is a protein that is not expressed on normal cells in the skin, lungs, salivary glands, pancreas, nor other tissues. In adenocarcinoma, the tumor cells produce too much labyrinthin causing them to express this protein on the surface of the tumor cells. One way to control the growth of these tumor cells is to teach the immune system to generate an immune response against the labyrinthin protein by vaccination against labyrinthin. GM-CSF, or sargramostim, is a protein that acts as a white blood cell growth factor. It has also been shown to stimulate immune system. Thus, administration of GM-CSF may help to boost the immune system response when given together with the vaccine. This study may improve the general knowledge about Labvax 3(22)-23 and how the body may generate an immune response to kill adenocarcinoma tumor cells. In the second phase of the study, participants will also receive pembrolizumab, which may improve anti-cancer activity when given with Labvax 3(22)-23 and GM-CSF.

DETAILED DESCRIPTION:
Phase 1: Up to 10 participants with advanced/ metastatic or recurrent adenocarcinoma of any primary site will be enrolled. Participants will be given LabVax 3(22)-23 (intradermally) and adjuvant GM-CSF (subcutaneously) on weeks 1, 2, 4, 8, and 12. Participants will be evaluated for 16 weeks, which include a follow-up exam 4 weeks after the last injection of vaccine or last injection, if injection(s) are stopped earlier. The study will be terminated if one death or two subjects have ≥3 adverse events that are at least possibly related to the study treatment. [Note: Phase 1 enrollment was completed as of December 2022]

Phase 2: Up to 67 participants with advanced/ metastatic or recurrent lung adenocarcinoma (Cohort A) or non-lung adenocarcinomas (Cohort B). Pembrolizumab will be given intravenously every 3 weeks for up to 12 cycles on Day 1 of Weeks 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 31, and 34. Subjects will be given LabVax 3(22)-23 (intradermally) and adjuvant GM-CSF (subcutaneously) on weeks 7, 8, 10, 14, and 18. Participants will receive study treatment over 34 weeks if tolerating the treatment without tumor progression; a safety follow-up visit will occur 30 days post-last dose of study treatment. The participant's chart will be reviewed for up to 12 months post-last dose of study treatment. The study will be terminated if safety is insufficient following the lead-in period or if response is insufficient in Cohort A following the first expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign an informed consent form.
2. Subjects of at least 18 years of age with histologically confirmed diagnosis of adenocarcinoma.
3. Subjects with advanced/metastatic or recurrent solid tumors, with measurable or non-measurable disease as determined by RECIST version 1.1 are eligible for participation.
4. For Phase 2, Cohort A, participants must have:

   1. Histologically confirmed diagnosis of labyrinthin-positive lung adenocarcinoma.
   2. Received at least one line of anti-PD-1 or anti-PD-L1 therapy for any stage of NSCLC. Anti-PD-1 or anti-PD-L1 may have been given alone or in combination with other therapy.
   3. Progressed on at least one line of therapy if participant has a known sensitizing mutation for which an FDA-approved targeted therapy for NSCLC exists (e.g., EGFR, ALK, ROS1, BRAF, RET, NTRK, and MET sensitizing mutations).
5. For Phase 2, all subjects must be candidates for pembrolizumab therapy.
6. Subjects can either have progressed, had no response, or intolerance to prior cancer therapy. Patients must have recovered from all clinically significant treatment-related toxicities to grade 1 or less, except chemotherapy-associated peripheral neuropathy (motor or sensory), or endocrine-related AE, in which recovery to ≤ Grade 2 is allowed. For endocrine-related AEs, physiological doses of replacement therapy (e.g., levothyroxine, insulin, hydrocortisone, or other replacement therapy for adrenal or pituitary insufficiency, etc.) are allowed.
7. No limit on prior lines of therapy for metastatic disease. Prior chemotherapy, immunotherapy (including pembrolizumab) or molecularly targeted therapy must have been completed at least 3 weeks prior to initiating study treatment. Prior palliative radiation must have been completed at least 2 weeks prior to initiating study treatment.
8. Subjects with known untreated, active brain and/or leptomeningeal metastases are excluded. Subjects with treated brain metastasis who are neurologically stable and off steroids for at least one week are eligible.
9. All subjects must have an ECOG performance status of 0-1. 10 All subjects must have a life expectancy of ≥ 6 months at the time of initiating study treatment.

11. Subjects must demonstrate adequate organ function as defined below:

* Absolute neutrophil count (ANC) ≥1,000 cells / μL
* Absolute lym75,000 cells/μL
* Creatinine clearance as calculated per Cockcroft-Gault or MDRD formula ≥30 mL/min
* Total bilirubin ≤ 1.5 X ULN or direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 ULN
* AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN or ≤ 5 X ULN for subjects with liver 12. Because the effects of the study treatment on the unborn fetus or nursing infant are unknown, pregnant and nursing women are ineligible. Women of childbearing age must have a negative urine or serum pregnancy test (HCG) within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

  13. Confirmation of adequate archival tumor specimens (i.e., sufficient specimens for ten, 5-7 µm thick, unstained sections).

Exclusion Criteria:

1. Subjects who have autoimmune diseases that require immunosuppressive medications other than prednisone ≤ 10 mg daily or equivalent. Physiological doses of replacement therapy (e.g., levothyroxine, insulin, hydrocortisone, or other replacement therapy for adrenal or pituitary insufficiency, etc.) are not considered a form of immunosuppressant and are allowed.
2. Subjects who have had a prior splenectomy are ineligible.
3. Pregnant or nursing women.
4. Any medical condition including additional malignancies, laboratory abnormalities, or psychiatric illness that in the opinion of the investigator would prevent the subject from participating and adhering to study related procedures.
5. Uncontrolled concomitant disease that in the opinion of the investigator would interfere with the subject's safety or compliance on trial.
6. Severe infection that in the opinion of the investigator would interfere with subject safety or compliance on trial within 4 weeks prior to enrollment.
7. Subjects who have contraindications to GM-CSF injections according to the package insert (e.g., subjects with excessive leukemic myeloid blasts in the bone marrow or peripheral blood (≥ 10%); known hypersensitivity to GM-CSF, yeast-derived products or any component of the product).

   Additional exclusion criteria for participants entering Phase 2:
8. Is receiving systemic steroid therapy (> 10 mg prednisone oral daily or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
9. Has a known history of active TB (Bacillus Tuberculosis)
10. Hypersensitivity to pembrolizumab or any of its excipients.
11. Has had a prior anti-cancer monoclonal antibody (mAb) within 3 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 3 weeks earlier.
12. Has had prior chemotherapy, targeted therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

    * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
    * Note: If subjects received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
13. Has known untreated, symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases requiring treatment, and are not using steroids (> 10 mg prednisone oral daily or equivalent) for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
14. Has known history of ≥ grade 3 pneumonitis or interstitial lung disease related to radiation, immunotherapy, chemotherapy, or targeted therapy.
15. Has an active infection requiring systemic therapy.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy.

    * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed. COVID vaccines are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose-limiting toxicities (DLT) | First LabVax 3(22)-23 injection through 14 days following the second LabVax 3(22)-23 injection
  Will be assessed according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (V)5.0. The type, grade, frequency and proportion of toxicities noted during the treatment period will be reported, along with associated 95% two-sided exact confidence interval of proportion. All adverse events noted by the investigator will be tabulated according to the affected body system.
Phase 1: Adverse events (AEs) | Up to 30 days after the last dose of study treatment
  Will be assessed according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (V)5.0. The type, grade, frequency and proportion of toxicities noted during the treatment period will be reported, along with associated 95% two-sided exact confidence interval of proportion. All adverse events noted by the investigator will be tabulated according to the affected body system.
Phase 2: Objective response rate (ORR) | Up to 12 months after last dose of study treatment
  Will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) version (V)1.1 guidelines. The fractions will be reported along with 95% two-sided exact confidence intervals. Comparisons between arms will be performed by Fisher's Exact tests. Investigators will also characterize the proportion who remain that either respond or have stable disease, compared to those who progress.

SECONDARY OUTCOMES:
Phase 1: Objective response rate (ORR) | Up to 12 months after last dose of study treatment
  Will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) version (V)1.1 guidelines. The fractions will be reported along with 95% two-sided exact confidence intervals. Comparisons between arms will be performed by Fisher's Exact tests. Investigators will also characterize the proportion who remain that either respond or have stable disease, compared to those who progress.
Phase 2: Dose-limiting toxicities (DLT) | Up to 30 days after the last LabVax 3(22)-23 vaccination
  Will be assessed according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (V)5.0. The type, grade, frequency and proportion of toxicities noted during the treatment period will be reported, along with associated 95% two-sided exact confidence interval of proportion. All adverse events noted by the investigator will be tabulated according to the affected body system.
Phase 2: Adverse events (AEs) | Up to 30 days after the last dose of study treatment
  Will be assessed according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (V)5.0. The type, grade, frequency and proportion of toxicities noted during the treatment period will be reported, along with associated 95% two-sided exact confidence interval of proportion. All adverse events noted by the investigator will be tabulated according to the affected body system.
Phase 2: Progression free survival (PFS) | Up to 12 months after last dose of study treatment
  PFS will be calculated as the time from initiation of immunotherapy to first documented evidence of disease progression or death, whichever comes first. Alive patients who have not been documented to have progression will be censored at the date of the latest clinical assessment that documented as being free of progression.
Phase 2: Overall survival (OS) | Up to 12 months after last dose of study treatment
  OS will be calculated as the time from diagnosis to death. Alive patients will be censored at the date of the latest follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Tianhong Li, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States

REFERENCES:
- [Result] Ma W, Zeng J, Montoya DJ, Toomey K, Zhou C, Chen S, Liu D, Babich M, Radosevich JA, Li T. Labyrinthin Expression Is Associated with Poor Prognosis in Patients with Non-Small-Cell Lung Cancer. Cancers (Basel). 2023 Feb 1;15(3):924. doi: 10.3390/cancers15030924. PMID 36765881